CLINICAL TRIAL: NCT01406665
Title: Assessment of Value of Skin Autofluorescence in Detecting Diabetes Mellitus or Impaired Glucose Tolerance. Comparison With Fasting Plasma Glucose and Glycated Hb
Brief Title: Skin Autofluorescence (AF) Decision Tree in Detecting Impaired Glucose Tolerance (IGT) or Diabetes Mellitus (DM)
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Prof. R.O.B. Gans, Head of Department Internal medicine, University medical Center Groningen Dept medicine
Other Study IDs: SAF-tree-IGTDM11; METc 2009-367 (Other: Institutional Review Board (IRB) UMCG)
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Diabetes Mellitus; Impaired Glucose Tolerance
Keywords: diabetes; impaired glucose tolerance
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — none retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- increased diabetes risk: the recruited group consists of persons with moderate to high risk for impaired glucose tolerance or diabetes

SUMMARY:
Early detection of (pre)diabetes, including impaired glucose tolerance is currently deficient because the best accepted standard, an oral glucose tolerance test (oGTT), is not feasible in a setting of screening or broad case-finding and other current methods lack in sensitivity. A previously reported study, and analysis of retrospective skin autofluorescence (AF) data, suggests that noninvasive skin AF may offer an alternative for detection of (pre)diabetes. The objective is to test the validity of a decision tree based on skin autofluorescence, and some simple clinical characteristics, as a detection tool for diabetes and impaired glucose tolerance. Sensitivity and specificity, positive and negative predictive value of this skin AF based decision model will be compared to those of fasting plasma glucose (FPG), glycated haemoglobin (HbA1c), and to two short questionnaires (Finnish Findrisk, and Cambridge score).

Study design: Skin AF, HbA1c and an oGTT (including an FPG) will be simultaneously performed in at least 120 persons with the characteristics described in the following paragraph. A Findrisk and Cambridge questionnaire will also be collected.

ELIGIBILITY:
Inclusion Criteria: -age >20 years

* additionally a priori intermediate risk for IGT/diabetes: by having at least one criterion from the metabolic syndrome, or by at least once having had an increased glucose or glycated hemoglobin value in the preceding two years, but these outside the range of diabetes/IGT

Exclusion Criteria:-known diabetes mellitus

* use of oral antidiabetics for other purposes than diabetes such as hepatic steatosis
* local skin disease of the lower arm obviating skin autofluorescence measurement
* known serious renal insufficiency (s-creatinine > 180 umol/l).
* inability to fill in questionnaires

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects identified from an outpatient (vascular, lipid) hospital-based group, with an intermediate risk of (pre)diabetes, as defined by an age >35 years, and additionally at least one criterion from the metabolic syndrome, or at least once an increased glucose or HbA1c value in the preceding two years, but these outside the range of diabetes/IGT
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
oGTT (WHO criteria)-defined impaired glucose tolerance or diabetes | individually immediately following test, for study <26 weeks
  numbers of true and false positives and negatives for oGTT (WHO criteria)-defined impaired glucose tolerance or diabetes are scored for Skin autofluorescence (based decision tree), FPG and HbA1c

SECONDARY OUTCOMES:
Findrisk diabetes questionnaire score | individually immediately after test, for study <26 weeks
  Findrisk diabetes questionnaire score is based on anthropometric data and questionnaire.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Gelre Ziekenhuis, Apeldoorn, Gelderland
  - University Medical Center Groningen, Groningen, Provincie Groningen